CLINICAL TRIAL: NCT04590950
Title: Monitoring and Pharmacodynamics Effect of Recombinant Factor IX Fc in Severe Haemophilia B Patients: a Real-life Study
Brief Title: Dosage and PD Study of Eftrenonacog-alfa
Acronym: BIOPAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191124
Record Dates: First submitted 2020-07-08; First posted 2020-10-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Severe Haemophilia B
Keywords: Chromogenic assay; Extended half-life product; Fc fusion protein; One-stage clotting assay; Pharmacodynamics
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Citrated plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single-group study: Severe haemophilia B patients substituted with eftrenonacog-alfa
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
The purpose of this study is to evaluate the performance of different methods for measuring factor IX activity levels in haemophilia B patients treated with eftrenonacog-alfa and assess its pharmacodynamics (PD) in a real-life setting.

DETAILED DESCRIPTION:
A recent European survey showed that increasing number of hemophilia B patients was switched from standard to extended half-life drugs. While some clinicians currently prefer to treat empirically rather than based on laboratory results, adoption of replacement therapy based on extended half-life products such as eftrenonacog-alfa may increase the interest in individualized pharmacokinetic assessments allowing the development of an initial dosing regimen. Thus inaccurate FIX activity measurements might be critical, especially when FIX trough level is used to tailor patient dosing regimens. It is therefore important that FIX activity levels are accurately determined allowing adequate recovery without increasing the cost of medical management of hemophilia B patients due to unnecessary dose corrections.

With the expansion of the prescription of eftrenonacog-alfa, the problem of accurately measuring its recovery has risen within hemostasis laboratories. Chronometric one-stage assays (OSA) are currently the most widely performed tests for FIX activity measurement. They are based on activated partial thromboplastin time (aPTT) reagent and factor-deficient plasma. Various aPTT reagents are commercialized. They could lead to a substantial variability in FIX results. Chromogenic two-stage assays (CSA) are less frequently used in clinical laboratories. They present fewer reagent choice compared to OSA. Several studies have evaluated OSA and CSA performances in samples spiked with eftrenonacog-alfa and have evidenced that some commonly used aPTT reagents would not be suitable for accurately monitoring this product. Whether these results are commutable to post-infusion samples collected from real-life patients remains unclear.

Unlike the measurement of a unique coagulation factor activity, thrombin generation assay (TGA) is a dynamic global test that explores the coagulation cascade as well as the anticoagulant pathways. TGA could be therefore a valuable tool to monitor replacement therapy in hemophilia B patients.

Hence the investigators sought in a real-life setting to compare 2 CSA and 1 OSA reagents to a product specific OSA in severe hemophilia B patients supplemented with eftrenonacog-alfa. The investigators also aimed to evaluate the pharmacodynamics (PD) of eftrenonacog-alfa using TGA.

ELIGIBILITY:
Inclusion Criteria:

* severe haemophilia B patients
* treated with eftrenonacog-alfa

Exclusion Criteria:

* any other haemostatic or replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe haemophilia B patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
FIX activity levels | One month
  2 chromogenic assays (Bio phen FIX and Rox FIX) and 2 chronometric assays (CK Prest with standard human plasma or FIX deficient plasma supplemented with eftrenonacog-alfa as calibrators)

SECONDARY OUTCOMES:
Thrombin generation assay | One month
  Thrombin generation assay is performed using a microplate fluorometer. Plasma samples are run using 20 μL low phospholipids reagent (PPP-reagent) (1 μM tissue factor and 4 micromoles (μM )phospholipid vesicles) or 20 μL Thrombin Calibrator. Assay is initiated by auto dispensing 20 μL of Fluo-Substrate solution containing calcium ions and fluorogenic substrate, Z-Gly-Gly-Arg-7-amino-4-methylcoumarin. Generated thrombin cleaves the substrate and fluorescence increase is monitored at 37 °C for 60 min with a measurement every 20 seconds.
  Thrombin scope®, version 5.0.0.742 is used to calculate the amount of thrombin generated over time taking into account for each sample the calibrator activity. Consequently, five parameters are reported by the Thrombin scope® the fist is lag time (LT; in min)
Thrombin generation assay | One month
  microplate fluorometer, time to peak
Thrombin generation assay | One month
  microplate fluorometer, peak height
Thrombin generation assay | One month
  microplate fluorometer, endogenous thrombin potential
Thrombin generation assay | One month
  microplate fluorometer, velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie biologique - Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peyvandi F, Garagiola I, Boscarino M, Ryan A, Hermans C, Makris M. Real-life experience in switching to new extended half-life products at European haemophilia centres. Haemophilia. 2019 Nov;25(6):946-952. doi: 10.1111/hae.13834. Epub 2019 Aug 16. PMID 31418967
- [Background] Sommer JM, Buyue Y, Bardan S, Peters RT, Jiang H, Kamphaus GD, Gray E, Pierce GF. Comparative field study: impact of laboratory assay variability on the assessment of recombinant factor IX Fc fusion protein (rFIXFc) activity. Thromb Haemost. 2014 Nov;112(5):932-40. doi: 10.1160/TH13-11-0971. Epub 2014 Aug 21. PMID 25144892
- [Background] Kitchen S, Tiefenbacher S, Gosselin R. Factor Activity Assays for Monitoring Extended Half-Life FVIII and Factor IX Replacement Therapies. Semin Thromb Hemost. 2017 Apr;43(3):331-337. doi: 10.1055/s-0037-1598058. Epub 2017 Mar 6. PMID 28264199
- [Background] Dargaud Y, Beguin S, Lienhart A, Al Dieri R, Trzeciak C, Bordet JC, Hemker HC, Negrier C. Evaluation of thrombin generating capacity in plasma from patients with haemophilia A and B. Thromb Haemost. 2005 Mar;93(3):475-80. doi: 10.1160/TH04-10-0706. PMID 15735797
- [Background] Bowyer AE, Shepherd MF, Kitchen S, Maclean RM, Makris M. Measurement of extended half-life recombinant factor IX products in clinical practice. Int J Lab Hematol. 2019 Apr;41(2):e46-e49. doi: 10.1111/ijlh.12953. Epub 2018 Dec 7. No abstract available. PMID 30536630
- [Background] Collins PW, Fischer K, Morfini M, Blanchette VS, Bjorkman S; International Prophylaxis Study Group Pharmacokinetics Expert Working Group. Implications of coagulation factor VIII and IX pharmacokinetics in the prophylactic treatment of haemophilia. Haemophilia. 2011 Jan;17(1):2-10. doi: 10.1111/j.1365-2516.2010.02370.x. Epub 2010 Aug 22. PMID 20731726
- [Background] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Background] Atsou S, Furlan F, Duchemin J, Ellouze S, Sourdeau E, Launois A, Roussel-Robert V, Stieltjes N, Combe S, Fontenay M, Curis E, Jourdi G. Pharmacodynamics of eftrenonacog-alfa (rFIX-Fc) in severe hemophilia B patients: A real-life study. Eur J Pharmacol. 2021 Jan 15;891:173764. doi: 10.1016/j.ejphar.2020.173764. Epub 2020 Nov 27. PMID 33249076